CLINICAL TRIAL: NCT07360795
Title: Do We Really Bleed in Percutaneous Nephrolithotomy? A Single-Surgeon, Single-Center Experience
Status: Completed | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Sponsor
Other Study IDs: FSCH-SB-2025-PCNL
Record Dates: First submitted 2026-01-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Urolithiasis
Keywords: Perkütan Nefrolitotomi; Clavien-Dindo Sınıflandırması; Kan Transfüzyonu
MeSH Terms: conditions — Urolithiasis | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous Nephrolithotomy (PCNL) Cohort: Patients who underwent percutaneous nephrolithotomy performed by a single surgeon at a single tertiary care center. This retrospective cohort includes patients whose perioperative and postoperative bleeding outcomes, transfusion requirements, and surgical complications were evaluated using existing medical records.
  Interventions: Procedure: Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous Nephrolithotomy — Percutaneous nephrolithotomy performed according to standard clinical practice for the treatment of renal calculi. All procedures were completed by a single experienced surgeon. No additional intervention, modification, or experimental procedure was applied as part of the study. Data related to perioperative and postoperative bleeding outcomes were collected retrospectively from existing medical records.

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is an effective and guideline-recommended surgical technique for the treatment of large and complex renal stones; however, perioperative bleeding remains one of its most significant complications. Reported bleeding and transfusion rates vary widely in the literature, potentially due to differences in surgical technique, surgeon experience, and institutional practices.

This retrospective, single-center study aims to evaluate perioperative and postoperative bleeding outcomes, transfusion requirements, and bleeding-related complications in patients who underwent PCNL performed by a single surgeon. The findings are intended to clarify whether the real-world bleeding risk associated with PCNL is lower than commonly reported.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is an effective and guideline-recommended surgical technique for the treatment of large and complex renal stones; however, perioperative bleeding remains one of its most significant complications. Reported bleeding and transfusion rates vary widely in the literature, potentially due to differences in surgical technique, surgeon experience, and institutional practices.

This retrospective, single-center study aims to evaluate perioperative and postoperative bleeding outcomes, transfusion requirements, and bleeding-related complications in patients who underwent PCNL performed by a single surgeon. The findings are intended to clarify whether the real-world bleeding risk associated with PCNL is lower than commonly reported. This is a retrospective, single-center observational study conducted at Elazığ Fethi Sekin City Hospital, Türkiye. Medical records of patients who underwent percutaneous nephrolithotomy between August 1, 2022, and December 20, 2025, will be reviewed retrospectively using the hospital information management system and anesthesia records.

All PCNL procedures were performed by a single experienced urologist using standardized surgical techniques. Demographic characteristics, perioperative variables, laboratory values, bleeding parameters, transfusion requirements, postoperative outcomes, and complications will be analyzed. Surgical complications will be classified according to the Clavien-Dindo classification system.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent percutaneous nephrolithotomy (PCNL)
* Availability of complete intraoperative and postoperative follow-up data
* Availability of preoperative and postoperative complete blood count and biochemical laboratory results

Exclusion Criteria:

* Pregnancy
* Conversion to open or laparoscopic surgery during PCNL
* Simultaneous additional surgical procedures, bilateral or synchronous bilateral PCNL
* Known coagulation disorders, hematological diseases, or active bleeding in the preoperative period
* Use of anticoagulant or antiplatelet therapy without appropriate perioperative management
* Preoperative blood transfusion requirement
* Severe intraoperative hemodynamic instability affecting the surgical course
* Missing hemoglobin or hematocrit data, insufficient transfusion or complication records
* Inadequate postoperative follow-up or transfer to another institutionConversion to open or laparoscopic surgery during PCNL
* Simultaneous additional surgical procedures, bilateral or synchronous bilateral PCNL
* Known coagulation disorders, hematological diseases, or active bleeding in the preoperative period
* Use of anticoagulant or antiplatelet therapy without appropriate perioperative management
* Preoperative blood transfusion requirement
* Severe intraoperative hemodynamic instability affecting the surgical course
* Missing hemoglobin or hematocrit data, insufficient transfusion or complication records
* Inadequate postoperative follow-up or transfer to another institution

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with nephrolithiasis who underwent percutaneous nephrolithotomy at a single tertiary care center. The study population consists of adult patients treated by a single surgeon, with perioperative and postoperative outcomes evaluated retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin Level | From the preoperative baseline to postoperative day 1 and throughout the length of hospital stay.
  The difference between preoperative and postoperative hemoglobin levels (g/dL) will be evaluated in patients undergoing percutaneous nephrolithotomy

SECONDARY OUTCOMES:
Change in Hematocrit Level | From the preoperative baseline to postoperative day 1 and throughout the length of hospital stay.
  The change in hematocrit (%) values between the preoperative and postoperative periods will be assessed
Estimated Intraoperative Blood Loss | During the surgical procedure.
  Estimated blood loss (mL) during percutaneous nephrolithotomy will be assessed based on intraoperative surgical records.
Postoperative Blood Transfusion Requirement | From postoperative day 1 until hospital discharge.
  The need for postoperative blood transfusion (yes/no) and the number of transfused packed red blood cell units will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No